CLINICAL TRIAL: NCT00952887
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of ACE-031 (ActRIIB-IgG1) in Healthy Postmenopausal Women
Brief Title: A Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of ACE-031 in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Richard Larouche, MD, Anapharm Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A031-02
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — ACVR2B protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACE-031 (Experimental): 8 dosing groups
  Interventions: Biological: ACE-031
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ACE-031 — Either 2 or 3 subcutaneous doses of ACE-031 over a period of one month, or 7 subcutaneous doses of ACE-031 over a period of 3 months.
  Other Names: ActRIIB-IgG1
  Arms: ACE-031
Biological: Placebo — Either 2 or 3 subcutaneous doses of placebo over a period of one month, or 7 subcutaneous doses of placebo over a period of 3 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish safe dose levels of ACE-031 in healthy postmenopausal women following multiple dose administration. This study will also evaluate if ACE-031 has an effect on muscle.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Body mass index (BMI) of ≥ 18.5 to < 32.

Exclusion Criteria:

* History of malignancy, except excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas
* History of clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease.
* History of opportunistic infection (e.g. invasive candidiasis or pneumocystis pneumonia) within 6 months prior to screening or serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening.
* Surgery within 3 months prior to Day 1 (other than minor cosmetic or dental procedures).
* Fever or symptomatic viral or bacterial infection within 7 days prior to Day 1.
* Donation or significant loss of blood within 2 months prior to Day 1.
* Hormone replacement therapy within 3 months prior to Day 1.
* Treatment with erythropoiesis stimulating agents (Epogen, Procrit, Aranesp, etc) within 2 months prior to Day 1.
* Systemic glucocorticoid therapy within 6 months prior to Day 1.
* Treatment with another investigational drug or approved therapy for investigational use within 1 month prior to Day 1.
* Previous treatment with ACE-031.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple, escalating doses of ACE-031 in healthy postmenopausal women | 6.5 months

SECONDARY OUTCOMES:
To estimate the pharmacokinetic (PK) and pharmacodynamic (PD) effects of multiple, escalating doses of ACE-031 | 6.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — Anapharm
Locations (2):
- Canada (2):
  - Acceleron Investigative Site, Montreal
  - Acceleron Investigative Site, Québec